CLINICAL TRIAL: NCT01255839
Title: A Prospective Multi-centre Randomised Comparison on Induction of Labour With Double-balloon Installation Device Versus Prostaglandin E2 Minprostin
Brief Title: The Balloon Project for Birth Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Henrik Nyholm, Department obstetrics and gynecology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-KA-01177-M
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2002-01

CONDITIONS: Induction Time; Apgar Score; Admission to Neonatal Unit; Vaginal Delivery; Caesarean Section
Keywords: double-balloon; balloon catheter; prostaglandin; minprostin; induction of labour; fetal outcome
MeSH Terms: interventions — Double-Balloon Enteroscopy; dinoprost tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Double-balloon (Active Comparator): The Double Balloon Catheter was applied (Atad 5) with 80 ml NaCl installed intrauterine above the intern orificium and 80 ml below in cervix/vagina.
  Interventions: Device: Double Balloon
- Prostglandin E2 (Active Comparator): The prostaglandin 2 minprostin (3mg) was applied vaginally
  Interventions: Drug: Minprostin

INTERVENTIONS:
Device: Double Balloon — The Double Balloon Catheter was applied (Atad 5) with 80 ml NaCl installed intrauterine above the intern orificium and 80 ml below in cervix/vagina.
  Arms: Double-balloon
Drug: Minprostin — The prostaglandin 2 minprostin (3mg) was applied vaginally
  Arms: Prostglandin E2

SUMMARY:
The use of prostaglandin E2 (PGE2) for induction of labour in women with unfavourable cervices is well-established1. There are, however, potential side effects to prostaglandins, in particular the risk of uterine hypertonicity which may affect fetal outcome. In theory a mechanical ripening based on dilatation of the cervix as well as induction of production of endogenous prostaglandin has potentially less influence on the fetal outcome but a Cochrane review from 2001 scrutinized studies on mechanical ripening versus placebo/no treatment or prostaglandin E2. They conclude there is insufficient data to evaluate the effectiveness in terms of likelihood of vaginal delivery in 24 hours, and emphasise the need for large sample size studies and substantive outcomes. Two later randomised studies compared mechanical ripening to PGE2 and found discrepant results regarding time from induction to delivery.

The primary purpose of the present study was in a randomized design to compare the efficacy of double-balloon catheter versus vaginal PGE2 (minprostin 3 mg) on induction of labour, duration of birth and fetal outcome. Secondary analyses were to evaluate the results for various subgroups, i.e. primipara/multipara, gemelli, vaginal birth after caesarean, preterm birth and intra uterine growth restriction.

DETAILED DESCRIPTION:
The study was a multicenter randomized study conducted at 7 labour yards in Denmark (Glostrup, Hillerød, Svendborg, Rigshospitalet, Næstved, Frederiksberg and Hvidovre). Participants were included from December 11 2002 till September 29 2005 after approval from The Danish National Committee on Biomedical Research Ethics and the data legislation. All participants were included after written and oral informed consent.

Eligible for inclusion were pregnancies with intact fetal membranes, vertex position and unripe cervix (Bishop score < 6) who had usual indications for induction of labour, i.e. prolonged pregnancy, pre-eclampsia/ hyper-tension, placental insufficiency, diabetes mellitus and twins.

Women were excluded under the following circumstances: Spontaneous labour or rupture of membranes, placenta previa, acute fetal distress, specific infections vagina/cervix (GBS, condyloma, acute herpes), asthma, glaucoma and allergy to latex. The participants were randomised to treatment arm by 'telephonic automatic voice response system randomisation'.

Induction of labour methods The balloon group The Double Balloon Catheter was applied (Atad 5) with 80 ml NaCl installed intrauterine above the intern orificium and 80 ml below in cervix/vagina. The Balloon catheter was inserted in the evening (8-9 p.m.) if the Bishop-score was below 6, however if the score was above 6 or the insertion was impossible the participant was considered failure. The catheter was removed after 12 h (or before if needed). The labour induction was continued by amniotomy either directly or after 2 hours mobilisation and laxative or after additional 2 hours of intravenous syntocinon drip. If by then amniotomy was not possible the participant was considered failure. After amniotomy if necessary for progression of contractions intravenous oxytocin-drip was started for 2-3 hours (figure 1). If further induction was necessary the participant was considered failure.

The minprostin group The prostaglandin 2 minprostin (3mg) was applied vaginally in the morning the day of induction if Bishop score was 6 or below. After 4-5 hours a second minprostin was inserted if amniotomy was not possible. If the labour was not induced the first day the procedure it was repeated the following day. If labour was not established within 48 hours after the first minprostin the participant was considered failure.

ELIGIBILITY:
Inclusion Criteria:

* pregnancies with intact fetal membranes
* vertex position
* unripe cervix Bishop score < 6)
* usual indications for induction of labour, i.e. prolonged pregnancy, pre-eclampsia/ hyper-tension, placental insufficiency, diabetes mellitus and twins

Exclusion Criteria:

* Spontaneous labour or rupture of membranes
* placenta previa
* acute fetal distress
* specific infections vagina/cervix (GBS, condyloma, acute herpes)
* asthma
* glaucoma
* allergy to latex

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 825 (Actual)
Dates: Start 2002-12; Primary Completion 2005-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
success of induction of labour, duration of birth and fetal outcome | at birth
  The primary purpose of the present study was in a randomized design to compare the efficacy of double-balloon catheter versus vaginal PGE2 (minprostin 3 mg) .

SECONDARY OUTCOMES:
the results for various subgroups, i.e. primipara/multipara, gemelli, vaginal birth after caesarean, preterm birth and intra uterine growth restriction | at birth

CONTACTS AND LOCATIONS:
Locations (1):
- Glostrup University Hospital, Glostrup Municipality, Glostrup, Denmark